CLINICAL TRIAL: NCT01798732
Title: Effect of Selective Laser Trabeculoplasty on the Intraocular Pressure Nycthemeral Rhythm.
Brief Title: PIO Laser Sclerectomy IOP SLT Sclerectomy
Acronym: PIO laser SPNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012; 2010-A00932-37 (Other: ID RCB)
Record Dates: First submitted 2012-12-12; First posted 2013-02-26 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Primary Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selective laser trabeculoplasty (Tango Laser, Ellex) (Experimental): Patients treated with selective laser trabeculoplasty (Tango Laser, Ellex, Minneapolis, USA)
  Interventions: Procedure: Selective Laser Trabeculoplasty (Tango Laser, Ellex)

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty (Tango Laser, Ellex) — One session of selective laser trabeculoplasty with the following parameters (inferior half-circumference, 50 shots, 0.8 to 1.3 mJ)

SUMMARY:
The main objective of this study is to characterize the changes in IOP over 24 hours after selective trabeculoplasty SLT (before and 1 and 6 months after treatment, decreased IOP, type of rhythm, mesor, acrophase, amplitude). The secondary objective is to evaluate changes in ocular perfusion pressure (arterial pressure - IOP) and ocular blood flow in the optic nerve head after selective laser trabeculoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open-Angle Glaucoma
* IOP more than 21 mmHg
* Progression under maximal medical therapy
* aged more than 18 years

Exclusion Criteria:

* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
IOP change over 24 hours after selective trabeculoplasty SLT according to chronobiological data (decrease of IOP; type of 24h-IOP rhythm and 24h-PPm rhythm: MESOR, acrophase, bathyphase, amplitude and modeling) | Baseline and 6 months

SECONDARY OUTCOMES:
Changes in the rate of ocular perfusion pressure (arterial pressure - IOP) and ocular blood flow in the optic nerve head after SLT. | Baseline and 6 months
  * To find predictive factors 1 month before efficacy of the treatment (after 6 month). Efficacy is defined by a mean IOP decrease, at least 30%, with a smoothed pressure-peaks (decrease at least 40% of pressure changes)
  * To characterize changes of ocular blood flow parameters (optic nerve head; Volume, Velocity and Flow): 20% at least of increase.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul ROMANET, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Khayi H, Pepin JL, Geiser MH, Tonini M, Tamisier R, Renard E, Baguet JP, Levy P, Romanet JP, Chiquet C. Choroidal blood flow regulation after posture change or isometric exercise in men with obstructive sleep apnea syndrome. Invest Ophthalmol Vis Sci. 2011 Dec 16;52(13):9489-96. doi: 10.1167/iovs.11-7936. PMID 22025580